CLINICAL TRIAL: NCT02079909
Title: A Phase 2 Multi-center, Randomized, Double Blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of T-817MA in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety of T-817MA in Patients With Mild to Moderate Alzheimer's Disease (US202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FUJIFILM Toyama Chemical Co., Ltd. (Industry)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T817MAUS202
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Alzheimer's
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- T-817MA-H (Experimental): 224 mg T-817MA once daily for first 4 weeks and 448 mg T-817MA once daily for the following weeks.
  Interventions: Drug: T-817MA-H
- T-817MA-L (Experimental): 224 mg T-817MA once daily
  Interventions: Drug: T-817MA-L
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T-817MA-H — 224 mg or 448 mg T-817 MA once daily
  Arms: T-817MA-H
Drug: T-817MA-L — 224 mg T-817 MA once daily
  Arms: T-817MA-L
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the efficacy of T-817MA as measured by ADAS-cog and ADCS-CGIC.

The secondary objectives are:

* To evaluate the safety and tolerability of T-817MA measured by clinical safety laboratories, physical examinations, ECGs and solicitation of adverse events.
* To evaluate the efficacy of T-817MA as measured by ADCS-ADL, FAQ, Neuropsychiatric Inventory (NPI) and Mini-mental State Examination (MMSE).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (post-menopausal or surgically sterile)
* Patients with Mild to moderate Alzheimer's disease who are receiving donepezil (Aricept®) or rivastigmine transdermal system (Exelon® Patch), . Memantine (Namenda®) is allowed only when prescribed in combination with donepezil or rivastigmine transdermal system.
* Age 55 to 85 inclusive
* Patients must be living in the community
* Patients must have an eligible informant or study partner (caregiver)
* Patients and eligible informant or study partner (caregiver) must be able to read and understand English.
* Informed consent obtained from both the patient and the caregiver

Exclusion Criteria:

* Patients with clinically significant cardiac, hepatic or renal impairment
* Patient have a dementia not of the Alzheimer's type etc (According to the protocol)
* Patients who are taking any drug other than donepezil or rivastigmine transdermal system for Alzheimer's disease, including olal rivastigmine (Exelon®), galantamine (Razadyne®)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2014-03; Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - UCSD Comprehensive Alzheimer's Program, La Jolla, California
  - UC Irvine Medical Center, Orange, California
  - Geriatric and Adult Psychiatry, LCC, Hamden, Connecticut
  - Yale University, Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Georgetown University Clinical Research Unit, Washington D.C., District of Columbia
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - University of Miami Miller-School of Medicine, Miami, Florida
  - Scientific Clinical Research, Inc, North Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Meridien Research, Tampa, Florida
  - Neuro Trials Research, Inc, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Indiana Medical Research, Elkhart, Indiana
  - Indiana University Health Partners, Adult Neurology Clinic, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas/Clinical and Translational Science Unit, Fairway, Kansas
  - University of Kentucky Sanders-Brown Center on Aging Clinic, Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Acadia Hospital, Bangor, Maine
  - Boston University Alzheimer's Disease Center, Boston, Massachusetts
  - University of Michigan Health System/ Michigan Clinical Research Unit, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Bronson Neurobehvioral Health, Paw Paw, Michigan
  - University of Nebraska Medical Center(Geri Psych), Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Global Medical Institutes, LLC;Princeton Medical Institute, Princeton, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Alzheimer's Disease Research Center of Mount Sinai, New York, New York
  - Columbia University Medical Center Sergievsky Center Taub Institute, New York, New York
  - The Nathan S. Kline Instituite for Psychiatric Research, Orangeburg, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest University (WFU) School of Medicine, Winston-Salem, North Carolina
  - Case Western Reserve University/ University Hospitals Case Medical Center, Beachwood, Ohio
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Hospital at the University of Pennsylvania, Penn Memory Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Alzheimer Disease Research Center, Pittsburgh, Pennsylvania
  - Abington Neurological Associates, LTD., Willow Grove, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Vanderbilt University Medical Center -VUIIS, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Cary J. Kohlenberg MD., SC dba IPC Research, Waukesha, Wisconsin

REFERENCES:
- [Derived] Schneider LS, Thomas RG, Hendrix S, Rissman RA, Brewer JB, Salmon DP, Oltersdorf T, Okuda T, Feldman HH; Alzheimer's Disease Cooperative Study TCAD Study Group. Safety and Efficacy of Edonerpic Maleate for Patients With Mild to Moderate Alzheimer Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2019 Nov 1;76(11):1330-1339. doi: 10.1001/jamaneurol.2019.1868. PMID 31282954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T-817MA-H | T-817MA-L | Placebo
Started | 158 | 166 | 158
Completed | 120 | 117 | 140
Not Completed | 38 | 49 | 18
Not completed — Adverse Event | 23 | 23 | 7
Not completed — Withdrawal by Subject | 9 | 17 | 4
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Death | 2 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Relocation etc. | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The overall numbers of baseline participants display patient numbers in the mITT population, the primary analysis population. The mITT population excludes patients who did not take any study drug or did not perform any efficacy evaluation post-baseline. Thus, the numbers are slightly difference from the ones in the participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | T-817MA-H | T-817MA-L | Placebo | Total
Number analyzed (Participants) | 154 | 159 | 156 | 469
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (7.8) | 71.9 (8.2) | 71.8 (7.5) | 71.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 81 | 89 | 252
  Male | 72 | 78 | 67 | 217
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 8 | 7 | 11 | 26
  White | 140 | 146 | 142 | 428
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 0 | 3
ApoE4 genotype [Count of Participants; unit: Participants]
  Non-carriers | 54 | 57 | 50 | 161
  Heterozygotes | 55 | 74 | 71 | 200
  Homozygotes | 32 | 21 | 27 | 80
  Unknown | 13 | 7 | 8 | 28
MMSE [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental Scale Examination (MMSE) is a validated, brief, frequently used screening instrument for Alzheimer's disease drug studies. The MMSE scale evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two overlapping pentagons. The MMSE is scored as the number of correctly completed items with a lower score indicative of poorer performance and greater cognitive impairment. The total score ranges from 0 (worse) to 30 (perfect performance).
  units on a scale | 18.4 (3.9) | 18.2 (3.8) | 18.2 (3.8) | 18.3 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: ADAS-cog Change From Baseline to Week 52
Description: The ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale) is a structured scale that evaluates memory (word recall, word recognition), reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). Ratings of spoken language, language comprehension, word finding difficulty, and ability to remember test instructions are also obtained. The test is scored in terms of errors, with higher scores reflecting poorer performance and greater impairment. Scores can range from 0 (best) to 70 (worse).
Time Frame: Baseline and 52 weeks
Population: The overall number of participants display the numbers of patients who were included in the mITT population and had baseline and at least one post-baseline ADAS-cog evaluation.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | T-817MA-H | T-817MA-L | Placebo
Number analyzed (Participants) | 117 | 115 | 137
units on a scale | 7.08 (0.756) | 7.45 (0.756) | 7.91 (0.727)
Statistical Analysis 1: Comparison: T-817MA-H vs Placebo; Test type: Superiority; p = 0.3919, Mixed Models Analysis; Mean Difference (Final Values) = -0.84

2. Primary Outcome: CGIC
Description: The ADCS-CGIC (Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change) is a validated categorical measure of change in the patient's clinical condition between baseline and follow-up visits. It measures whether the effects of active treatment are substantial enough to be detected by a skilled and experienced clinician on the basis of a clinical interview and examination. It relies on both direct examination of the patient and an interview of the study partner. A skilled and experienced clinician who is blinded to treatment assignment rates the patient on a 7-point Likert scale, ranging from 1 (marked improvement) to 7 (marked worsening). It is suggested that the instrument has distinct clinical utility in assessing change in AD clinical trials.
Time Frame: 52 weeks
Population: The overall number of participants display the numbers of patients who were included in the mITT population and had at least one post-baseline CGIC evaluation.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | T-817MA-H | T-817MA-L | Placebo
Number analyzed (Participants) | 118 | 116 | 138
units on a scale | 5.25 (0.1) | 5.24 (0.1) | 5.22 (0.1)
Statistical Analysis 1: Comparison: T-817MA-H vs Placebo; Test type: Superiority; p = 0.7588, Mixed Models Analysis; Mean Difference (Final Values) = 0.04

3. Secondary Outcome: ADCS-ADL Change From Baseline to Week 52
Description: The ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living) is a validated tool for assessing instrumental and basic activities of daily living based on a 23-item structured interview of the study partner. The scale has a range of 0 to 78, with lower scores indicating greater impairment.
Time Frame: Baseline and 52 weeks
Population: The overall number of participants display the numbers of patients who were included in the mITT population and had baseline and at least one post-baseline ADCS-ADL evaluation.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | T-817MA-H | T-817MA-L | Placebo
Number analyzed (Participants) | 118 | 118 | 140
units on a scale | -10.01 (0.991) | -11.07 (0.992) | -11.29 (0.957)
Statistical Analysis 1: Comparison: T-817MA-H vs Placebo; Test type: Superiority; p = 0.3212, Mixed Models Analysis; Mean Difference (Final Values) = 1.29

ADVERSE EVENTS:
Time Frame: 52weeks
Arm/Group | T-817MA-H | T-817MA-L | Placebo
All-Cause Mortality (participants affected / at risk) | 2/158 | 2/166 | 0/158
Serious Adverse Events (participants affected / at risk) | 26/158 | 25/166 | 20/158
Other Adverse Events (participants affected / at risk) | 132/158 | 133/166 | 119/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-817MA-H (N=158) | T-817MA-L (N=166) | Placebo (N=158)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1 | 1
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia Influenzal (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Altered State of Consciousness (Nervous system disorders) | 0 | 0 | 1
Cerebral Haematoma (Nervous system disorders) | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 3
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0
Abnormal Behaviour (Psychiatric disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 1 | 0
Delirium (Psychiatric disorders) | 3 | 1 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T-817MA-H (N=158) | T-817MA-L (N=166) | Placebo (N=158)
Nasopharyngitis (Infections and infestations) | 4 | 4 | 9
Urinary tract infection (Infections and infestations) | 21 | 17 | 22
Agitation (Psychiatric disorders) | 4 | 5 | 14
Anxiety (Psychiatric disorders) | 7 | 9 | 12
Depression (Psychiatric disorders) | 8 | 6 | 7
Dizziness (Nervous system disorders) | 11 | 7 | 3
Headache (Nervous system disorders) | 9 | 16 | 10
Diarrhoea (Gastrointestinal disorders) | 49 | 34 | 20
Nausea (Gastrointestinal disorders) | 9 | 13 | 6
Vomiting (Gastrointestinal disorders) | 9 | 8 | 7
Weight decreased (Investigations) | 8 | 4 | 3
Fall (Injury, poisoning and procedural complications) | 12 | 14 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02079909/Prot_SAP_000.pdf